CLINICAL TRIAL: NCT02077673
Title: Robotic Assisted Laparoscopy Versus Open Gastroesophageal Resection; Effects on the Mesenteric Traction Reflex and PGI2 Levels
Brief Title: Gastric Microperfusion in Patients Undergoing Gastroesophageal Resections
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Rikard Ambrus, MD, Rigshospitalet, Denmark
Other Study IDs: H-2-2013-101; 30-1152 (Registry Identifier: The Danish Data Protection Agency)
Record Dates: First submitted 2014-02-12; First posted 2014-03-04 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Surgery
Keywords: GEJ-cancer; surgery; gastroesophageal resection; gastroesophageal anastomosis; anastomotic leakage
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples Without DNA — Serum Tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- open surgery: 25 patients undergoing open gastroesophageal resection
- robotic-assissted surgery: 25 patients under-going robotic-assisted gastroesophageal surgery

SUMMARY:
Gastroesophageal resection because of gastroesophageal junction (GEJ) adenocarcinoma is a massive surgical intervention. Currently, gastroesophageal cancer surgery is performed with upper laparotomy followed by thoracotomy at the Department of Surgical Gastroenterology, Rigshospitalet, Denmark. However, minimal invasive techniques (MIT), e.g. robotic assisted laparoscopy, is in the progress of being implemented in this field as they are hypothesized to be more beneficial for the patients, and in some aspects better than conventional laparoscopic surgery.

The operative procedure is often complicated by low blood pressure (systolic blood pressure less than 90 mm Hg is experienced in more than 30 % of the patients) and is probably accompanied by a reduced splanchnic microcirculatory flow, leading to increased morbidity. Hypotension may be due to several factors, among them are epidural analgesia, mesentery traction reflex, and inflammatory and vasoactive hormones.

Aim of the project

The aim of the project is, through a series of sub-projects, to validate or invalidate the relationship between changes in the microcirculatory blood flow in the stomach and the systemic hemodynamic changes. Furthermore, the aim is to assess the changes in the microcirculatory blood flow as a consequence of the thoracic epidural anesthesia. In addition, the aim is to assess the hypothesis that the mesenteric traction reflex and changes in the PGI2 levels may influence systemic hemodynamic changes, and that robotic assisted MIT will attenuate the mesenteric traction reflex and changes in PGI2 compared to open surgery.

DETAILED DESCRIPTION:
Background:

Gastroesophageal resection because of gastroesophageal junction (GEJ) adenocarcinoma is a massive surgical intervention. Nevertheless, surgery is the only treatment with significant long-term survival. Currently, gastroesophageal cancer surgery is performed with upper laparotomy followed by thoracotomy at the Department of Surgical Gastroenterology, Rigshospitalet, Denmark. However, minimal invasive techniques (MIT), e.g. robotic assisted laparoscopy, is in the progress of being implemented in this field as they are hypothesized to be more beneficial for the patients, and in some aspects better than conventional laparoscopic surgery [1]. The benefits of MIT are believed to be due to several factors, a smaller surgical stress response [2] and less pain [3] resulting in earlier mobilization, to mention a few.

When reconstructing the gastrointestinal continuity, a gastric tube is prepared from the upper part of the remaining stomach. It is challenging to visualize, if the remaining stomach has adequate blood supply. Earlier studies have shown an up to 70 % reduction in blood flow, to the upper part of the remnant stomach [4-6], and ischemia is one of the most significant causes of anastomotic leakage [7, 8]. Anastomotic leakage occurs in up to 10 % of the patients and is fatal in up to 50 %. Furthermore, a recent study originated from the investigators department demonstrated, that patients experiencing anastomotic leakage after gastroesophageal cancer resection, have a significantly reduced long-term survival, even when early death and other postoperative complications were accounted for [9]. The overall 5-year survival rates in patients with and without anastomotic leakage were 20 and 35 %, respectively. Therefore, sufficient blood flow to the area of anastomosis is of paramount concern. Different techniques have been used in the attempt to assess the microcirculation during gastroesophageal resection [5, 10-13]. However, none of these techniques has proven to be practical, reliable, and time-efficient, and therefore not being routinely implemented in the clinical settings.

During open gastroesophageal resection, hypotension is common (systolic blood pressure less than 90 mm Hg is experienced in more than 30 % of the patients) and is probably accompanied by a reduced gastric microcirculatory flow. The hypotension may be due to several factors;

* Sympathic nerve system blockage due to thoracic epidural neuraxial anesthesia: Several studies have found reduced splanchnic flow after epidural anesthesia, which was associated with a decrease in systemic resistance and mean arterial pressure [14, 15]. The impact of the time-point for activation of epidural analgesia, on complications in the postoperative period is unknown. An unpublished study (Nielsen T: "Increased cardiac output after Whipple's procedure for pancreatic cancer") suggests that early activation during operation leads to significantly longer stay in the recovery ward after the surgery.
* The initial manipulation of viscera, results in a mesenteric traction reflex (also called eventration syndrome) with vasodilatation and secondary hypotension [16, 17]. The reason for mesenteric traction reflex is unknown, but is believed to be elicited by traction on the mesenterial blood vessels, resulting in a local release of prostacyclin (PGI2) from the endothelium. This reflex has mainly been shown to occur during pancreatic, gastric and aortic surgery, where manipulation of the mesenteric root is inevitable [18-21]. PGI2 is a potent vasodilatator, with inhibitory effect on platelet aggression and on vascular smooth cell proliferation [22-24].

Microcirculatory measurements:

Laser Speckle Contrast Imaging (LSCI) is a relatively new technique for microcirculatory monitoring. When laser light encounters a surface of an object, a random interference effect generates, called laser speckle contrast. The speckle pattern changes depending on the velocity of the object, and it is possible to get information regarding the object's movements, by the fluctuations in the speckle pattern. By measuring the concentration and velocity of blood cells, tissue perfusion may be assessed by LSCI technique. A real-time and non-touch measurement can be made on a large field (0.5 cm x 0.7 cm up to 15 cm x 20 cm). The camera is placed at a distance of 20-30 cm and measures the relative flow (flux) in the regions of interest. The measurement is at a depth of 1-2 mm by infrared light reflected from circulating erythrocytes in the micro-vessels.

Hypothesis and aim:

Robot-assisted laparoscopic surgery alters the hemodynamics and microcirculation in the splanchnic system by reduced release of vasoactive substances, such as PGI2, compared to open surgery. With this study, the investigators wish to evaluate hemodynamic fluctuations and gastric microcirculation, and correlate these to serum levels of PGI2 at different stages of surgery in robotic assisted laparoscopic surgery and open surgery, respectively.

Methods:

2 × 25 consecutive patients selected for robotic assisted laparoscopic or open surgery. Hemodynamic assessments are according to standardized methods. Blood samples will be drawn at: 1) after induction of anesthesia, 2) when the peritoneum is first entered, 3) after 15 min. of surgery, 4) after liberation of stomach, 5) after abdominal skin closure, 6) after extraction of the gastric conduit into the thorax, 7) after formation of the anastomosis, 8) after thoracic skin closure, 9) 18 hours after surgery. LSCI will be used to measure the microcirculation at two locations (3 cm from the pylorus and just below the site of the anastomosis (the body)) on the stomach five times during open surgery, and twice during the thoracic part of robotic assisted laparoscopic surgery.

Statistics:

Statistical power-calculation is carried out on an expected difference of the occurrence of mesenteric traction reflex between patients operated with open vs. MIT. By using sample size of 50 comparing percentages where group one is 55 % and group two is 12 % [17], a requirement of 18 patients in each group is calculated in order to obtain a statistical power greater than 0.80 with a α-level of <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with adenocarcinoma in the gastroesophageal junction
* Patients assumed to be resectable

Exclusion Criteria:

* lack of consent
* non-adenocarcinomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited at; The Department of Surgical Gastroenterology, Rigshospitalet, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
the occurence of anastomotic leakage | 7 days post-operative
  Anastomotic insufficiency is defined as leakage identified by:
  1. X-ray of the esophagus with water-soluble contrast on the 7.th day after operation, or
  2. CT-scan because of clinical signs (e.g. fever, pain), or
  3. Gastroscopy in critically ill patients.

SECONDARY OUTCOMES:
The occurrence of Mesenteric Traction Reflex | the initial 60 minutes of surgery
  The occurrence of Mesenteric Traction Reflex is defined as:
  1. A decrease in systemic vascular resistance (SVR) of more than 20 % and / or 900 dyne • s • cm-5 in relation with surgery of the stomach
  2. A decrease in systolic blood pressure of more than 20 %
  3. Measurable increase of the release of PGI2 in relation to decreased SVR and blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bo Svendsen, prof., MD, Study Director — Rigshospitalet, Denmark; Michael P Achiam, MD, PhD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Department of Surgical Gastroenterology, Rigshospitalet, Copenhagen Ø, Denmark

REFERENCES:
- [Background] Daouadi M, Zureikat AH, Zenati MS, Choudry H, Tsung A, Bartlett DL, Hughes SJ, Lee KK, Moser AJ, Zeh HJ. Robot-assisted minimally invasive distal pancreatectomy is superior to the laparoscopic technique. Ann Surg. 2013 Jan;257(1):128-32. doi: 10.1097/SLA.0b013e31825fff08. PMID 22868357
- [Background] Braga M, Vignali A, Zuliani W, Radaelli G, Gianotti L, Martani C, Toussoun G, Di Carlo V. Metabolic and functional results after laparoscopic colorectal surgery: a randomized, controlled trial. Dis Colon Rectum. 2002 Aug;45(8):1070-7. doi: 10.1007/s10350-004-6362-2. PMID 12195192
- [Background] Gramigni E, Bracco D, Carli F. Epidural analgesia and postoperative orthostatic haemodynamic changes: observational study. Eur J Anaesthesiol. 2013 Jul;30(7):398-404. doi: 10.1097/EJA.0b013e32835b162c. PMID 23435278
- [Background] Briel JW, Tamhankar AP, Hagen JA, DeMeester SR, Johansson J, Choustoulakis E, Peters JH, Bremner CG, DeMeester TR. Prevalence and risk factors for ischemia, leak, and stricture of esophageal anastomosis: gastric pull-up versus colon interposition. J Am Coll Surg. 2004 Apr;198(4):536-41; discussion 541-2. doi: 10.1016/j.jamcollsurg.2003.11.026. PMID 15051003
- [Background] Gomes M, Ramacciotti E, Miranda F Jr, Henriques AC, Fagundes DJ. Vascular flow of the gastric fundus after arterial devascularization: an experimental study. J Surg Res. 2009 Mar;152(1):128-34. doi: 10.1016/j.jss.2008.04.016. Epub 2008 May 7. PMID 18805545
- [Background] Thomas DM, Langford RM, Russell RC, Le Quesne LP. The anatomical basis for gastric mobilization in total oesophagectomy. Br J Surg. 1979 Apr;66(4):230-3. doi: 10.1002/bjs.1800660404. PMID 454988
- [Background] Pacheco PE, Hill SM, Henriques SM, Paulsen JK, Anderson RC. The novel use of intraoperative laser-induced fluorescence of indocyanine green tissue angiography for evaluation of the gastric conduit in esophageal reconstructive surgery. Am J Surg. 2013 Mar;205(3):349-52; discussion 352-3. doi: 10.1016/j.amjsurg.2012.11.005. PMID 23414958
- [Background] Reavis KM. The esophageal anastomosis: how improving blood supply affects leak rate. J Gastrointest Surg. 2009 Sep;13(9):1558-60. doi: 10.1007/s11605-009-0906-7. Epub 2009 May 5. No abstract available. PMID 19415398
- [Background] Kofoed SC, Calatayud D, Jensen LS, Jensen MV, Svendsen LB. Intrathoracic anastomotic leakage after gastroesophageal cancer resection is associated with reduced long-term survival. World J Surg. 2014 Jan;38(1):114-9. doi: 10.1007/s00268-013-2245-9. PMID 24129798
- [Background] Boyle NH, Pearce A, Hunter D, Owen WJ, Mason RC. Scanning laser Doppler flowmetry and intraluminal recirculating gas tonometry in the assessment of gastric and jejunal perfusion during oesophageal resection. Br J Surg. 1998 Oct;85(10):1407-11. doi: 10.1046/j.1365-2168.1998.00943.x. PMID 9782026
- [Background] Murawa D, Hunerbein M, Spychala A, Nowaczyk P, Polom K, Murawa P. Indocyanine green angiography for evaluation of gastric conduit perfusion during esophagectomy--first experience. Acta Chir Belg. 2012 Jul-Aug;112(4):275-80. PMID 23008991
- [Background] Schilling MK, Redaelli C, Maurer C, Friess H, Buchler MW. Gastric microcirculatory changes during gastric tube formation: assessment with laser Doppler flowmetry. J Surg Res. 1996 Apr;62(1):125-9. doi: 10.1006/jsre.1996.0184. PMID 8606499
- [Background] Schroder W, Beckurts KT, Stahler D, Stutzer H, Fischer JH, Holscher AH. Microcirculatory changes associated with gastric tube formation in the pig. Eur Surg Res. 2002 Nov-Dec;34(6):411-7. doi: 10.1159/000065709. PMID 12403940
- [Background] Gould TH, Grace K, Thorne G, Thomas M. Effect of thoracic epidural anaesthesia on colonic blood flow. Br J Anaesth. 2002 Sep;89(3):446-51. PMID 12402724
- [Background] Lundberg J, Lundberg D, Norgren L, Ribbe E, Thorne J, Werner O. Intestinal hemodynamics during laparotomy: effects of thoracic epidural anesthesia and dopamine in humans. Anesth Analg. 1990 Jul;71(1):9-15. doi: 10.1213/00000539-199007000-00002. PMID 2194404
- [Background] Brinkmann A, Seeling W, Wolf CF, Kneitinger E, Junger S, Rockemann M, Oettinger W, Georgieff M. [The effect of thoracic epidural anesthesia on the pathophysiology of the eventration syndrome]. Anaesthesist. 1994 Apr;43(4):235-44. doi: 10.1007/s001010050053. German. PMID 8179173
- [Background] Nomura Y, Funai Y, Fujimoto Y, Hori N, Hirakawa K, Hotta A, Nakamoto A, Yoshikawa N, Ohira N, Tatekawa S. Remifentanil increases the incidence of mesenteric traction syndrome: preliminary randomized controlled trial. J Anesth. 2010 Oct;24(5):669-74. doi: 10.1007/s00540-010-0998-y. Epub 2010 Aug 7. PMID 20694481
- [Background] Brinkmann A, Seeling W, Rockemann M, Junge JH, Radermacher P, Wiedeck H, Buchler MW, Georgieff M. Changes in gastric intramucosal pH following mesenteric traction in patients undergoing pancreas surgery. Dig Surg. 1999;16(2):117-24. doi: 10.1159/000018703. PMID 10207237
- [Background] Bucher M, Kees FK, Messmann B, Lunz D, Rath S, Zelenka M, Schlitt HJ, Hobbhahn J. Prostaglandin I2 release following mesenteric traction during abdominal surgery is mediated by cyclooxygenase-1. Eur J Pharmacol. 2006 May 1;536(3):296-300. doi: 10.1016/j.ejphar.2006.03.009. Epub 2006 Mar 13. PMID 16581062
- [Background] Gottlieb A, Skrinska VA, O'Hara P, Boutros AR, Melia M, Beck GJ. The role of prostacyclin in the mesenteric traction syndrome during anesthesia for abdominal aortic reconstructive surgery. Ann Surg. 1989 Mar;209(3):363-7. doi: 10.1097/00000658-198903000-00018. PMID 2647052
- [Background] Hudson JC, Wurm WH, O'Donnel TF Jr, Kane FR, Mackey WC, Su YF, Watkins WD. Ibuprofen pretreatment inhibits prostacyclin release during abdominal exploration in aortic surgery. Anesthesiology. 1990 Mar;72(3):443-9. doi: 10.1097/00000542-199003000-00009. PMID 2106806
- [Background] Kothapalli D, Stewart SA, Smyth EM, Azonobi I, Pure E, Assoian RK. Prostacylin receptor activation inhibits proliferation of aortic smooth muscle cells by regulating cAMP response element-binding protein- and pocket protein-dependent cyclin a gene expression. Mol Pharmacol. 2003 Aug;64(2):249-58. doi: 10.1124/mol.64.2.249. PMID 12869629
- [Background] Weksler BB, Marcus AJ, Jaffe EA. Synthesis of prostaglandin I2 (prostacyclin) by cultured human and bovine endothelial cells. Proc Natl Acad Sci U S A. 1977 Sep;74(9):3922-6. doi: 10.1073/pnas.74.9.3922. PMID 333448
- [Background] Wharton J, Davie N, Upton PD, Yacoub MH, Polak JM, Morrell NW. Prostacyclin analogues differentially inhibit growth of distal and proximal human pulmonary artery smooth muscle cells. Circulation. 2000 Dec 19;102(25):3130-6. doi: 10.1161/01.cir.102.25.3130. PMID 11120706
- [Derived] Strandby RB, Ambrus R, Secher NH, Goetze JP, Achiam MP, Svendsen LB. Plasma pro-atrial natriuretic peptide to estimate fluid balance during open and robot-assisted esophagectomy: a prospective observational study. BMC Anesthesiol. 2017 Feb 3;17(1):20. doi: 10.1186/s12871-017-0314-6. PMID 28159014